CLINICAL TRIAL: NCT04300465
Title: Evaluating the Effects of the MySláinte Community Lifestyle Intervention Program in Addressing Common Drivers of Disease in a Cohort of Chronic Disease Patients and Their Partners: a Pilot Study
Brief Title: MySlainte: Testing the Effect of Involving Partners in a CVD Prevention Community Lifestyle Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University of Ireland, Galway, Ireland (Other)
Responsible Party: Principal Investigator, Prof. John William McEvoy, Professor, National University of Ireland, Galway, Ireland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: C.A.2322
Record Dates: First submitted 2020-03-02; First posted 2020-03-09 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Rheumatoid Arthritis; Chronic Kidney Diseases; Cardiovascular Risk Factor; Partner, Domestic
Keywords: Rheumatoid Arthritis; Chronic Kidney Disease; Cardiovascular Risk Factors; Lifestyle Intervention; Chronic Disease
MeSH Terms: conditions — Arthritis, Rheumatoid; Renal Insufficiency, Chronic; Chronic Disease

STUDY DESIGN:
Intervention Model Description: Randomised parallel design. 2 study groups and within each group there are 2 arms.
  Patients with stable rheumatoid arthritis (RA) and their partners
  * 16 RA patients + 16 partners
  * each pairing is randomised into 1 of 2 groups
    1. With partner: The RA patients + their partners partake in the the intervention (8 RA patients and 8 partners)
    2. Without partner: the RA patients partake in the intervention alone (8 patients) The partner does not partake in the intervention (8 partners).
  Patients with stable stage 3 or 4 chronic kidney disease (CKD) and their partners
  * 16 CKD patients + 16 partners
  * each pairing is randomised into 1 of 2 groups
    1. With partner: The CKD patients and their partners partake in the the intervention (8 CKD patients and 8 partners)
    2. Without partner: the CKD patients partake in the intervention alone (8 patients). The partner does not partake in the intervention (8 partners)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Rheumatoid arthritis - With Partner Group (Experimental): In this group patients with stable rheumatoid arthritis and their partners both undergo an initial assessment, the 10 week intervention phase and then an end of program assessment together. The intervention phase includes weekly exercise classes, individualised exercise prescription, health promotion workshops, individualised goal setting and optimisation of cardioprotective medications.
  Interventions: Behavioral: 10 week MySlainte Program
- Rheumatoid arthritis - Without Partner Group (Active Comparator): In this group patients with stable rheumatoid arthritis undergo an initial assessment, the 10 week intervention phase and then the end of program assessment. Their partners attend the initial assessment and the end of program assessment but do not partake in the 10 week intervention phase. During the 10 week period these partners receive usual care from their GP's.
  For the patients with rheumatoid arthritis, the 10 week intervention phase includes weekly exercise classes, individualised exercise prescription, health promotion workshops, individualised goal setting and optimisation of cardioprotective medications.
  Interventions: Behavioral: 10 week MySlainte Program
- Chronic Kidney Disease - With Partner Group (Experimental): In this group patients with stable stage 3 or 4 chronic kidney disease and their partners both undergo an initial assessment, the 10 week intervention phase and then an end of program assessment together. The intervention phase includes weekly exercise classes, individualised exercise prescription, health promotion workshops, individualised goal setting and optimisation of cardioprotective medications.
  Interventions: Behavioral: 10 week MySlainte Program
- Chronic Kidney Disease - Without Partner Group (Active Comparator): In this group patients with stable stage 3 or 4 chronic kidney disease undergo an initial assessment, the 10 week intervention phase and then the end of program assessment. Their partners attend the initial assessment and the end of program assessment but do not partake in the 10 week intervention phase. During the 10 week period these partners receive usual care from their GP's.
  For the patients with chronic kidney disease, the 10 week intervention phase includes weekly exercise classes, individualised exercise prescription, health promotion workshops, individualised goal setting and optimisation of cardioprotective medications.
  Interventions: Behavioral: 10 week MySlainte Program

INTERVENTIONS:
Behavioral: 10 week MySlainte Program — The intervention consists of a 10 week community based lifestyle intervention program. It consists of a weekly 1 hour exercise class, a weekly 1 hour health promotion workshop as well as individualised goal setting, exercise prescription and optimisation of cardioprotective medications.
  This program is delivered by a multi-disciplinary team; including a physiotherapist, occupational therapist, dietitian, clinical nurse specialist and physician. It will be delivered through a registered Irish charity, Croí.

SUMMARY:
MySláinte is a 12-week community-based, multi-disciplinary preventive and lifestyle intervention program to reduce CVD risk factors. It includes weekly exercise classes with educational workshops on understanding lifestyle risk factors as well as optimisation of cardiovascular medications. It will be delivered by a multidisciplinary team including: a nurse, dietician, physiotherapist and physician and builds on the previously developed protocols of the successful MyAction program. The MySlainte study aims to expand on the MyAction program by looking at a broader range of patients with chronic disease who have suboptimal lifestyle drivers for many preventable diseases. Importantly, MySlainte also aims to assess if there is a difference in outcome between those who complete the program with their partner compared to those who complete the program alone.

DETAILED DESCRIPTION:
The prevalence of chronic diseases in Ireland is increasing and places significant burden both on the individual and family unit, but also on an already overstretched healthcare system. Many chronic diseases are preventable and frequently share common risk factor and unhealthy lifestyle profiles; which offers a unique opportunity to intervene, address and modify these common disease drivers, and potentially prevent disease complications.

The MyAction program and previous similar programs have successfully been run by Croí/NIPC (based in Galway, www.nipc.ie) in an effort to combat common cardiovascular risk factors. These programs have demonstrated that addressing and modifying risk factors is both effective and sustainable. Expanding programs like these to a broader group of chronic disease patients with overlapping modifiable risks could lead to multi-factorial benefits: prevention is better than cure. While cardiac and pulmonary rehab are well established programs, patients with other chronic diseases do not currently have access to such focused interventions in Galway. Chronic kidney disease and rheumatoid arthritis are two such chronic diseases that have a particularly high cardiovascular risk burden, and so may benefit from a focused intervention program.

Chronic kidney disease is a worldwide public health problem with an estimated prevalence of 11.8% in Ireland. With chronic kidney disease comes a myriad of other co-morbidities and increased rate of all-cause mortality. Significantly, cardiovascular disease is the primary contributor to increased morbidity and mortality in this patient cohort. In fact, in patients with Stage 3 CKD, the incidence of cardiovascular mortality is higher than the incidence of kidney failure. This makes prevention of drivers of cardiovascular disease a key component in managing these patients.

Lifestyle and exercise programs may have an even broader range of benefit in this patient group. Through inflammation, uremic toxins, and dysregulation of key proteins and hormones a second major consequence of CKD is sarcopenia and skeletal muscle dysfunction. This is compounded by the fact that physical activity in all stages of CKD are low, which leads to decreased quality of life, increased falls risk and associated morbidity. Previous programs have demonstrated the benefits of exercise in this group. The MySláinte program aims to build on this by tackling a broader range of modifiable risk factors.

Similarly, patients with rheumatoid arthritis have an increased risk of cardiovascular disease due to a complex interplay between systemic inflammation and a higher prevalence of traditional CVD risk factors. Despite recommendations by European League against Rheumatism (EULAR) of the importance of emphasising positive lifestyle choices, a recently published article by Malm concluded that discussions regarding lifestyle improvements (including exercise, smoking, drinking and diet) are suboptimal in these patients. Exercise programs have also been shown to be of benefit in these patient groups in decreasing falls rates, as well as improving health related quality of life measures.

It has previously been described that a concordance of behavioural risk factors exists between patients with coronary artery disease and their spouses. Similarly, spouses of patients with hypertension have increased odds of hypertension themselves. The same is seen in patients with type 2 diabetes, with spouses of patients with type 2 diabetes having a higher risk of developing type 2 diabetes. In keeping with that, it has been demonstrated that including both patients and their partners in lifestyle intervention programs improves not only the patients risk factor profile, but also that of the partners. It has also been suggested that couples who complete programs together may in fact do better than those who enter as individuals. Interestingly, even when lifestyle interventions are aimed only at a patient, spouses have shown to benefit indirectly from such programs in a knock on effect termed the "ripple effect". These concepts highlight the importance of considering a patient's support network when undergoing a lifestyle intervention. They also highlight a potentially unique opportunity to improve the lifestyles, and hence risk factor profiles, of entire households. Previously, the MyAction program had invited participants to bring their partners to the program. Unfortunately, due to funding issues, this part of the program was gradually phased out. However, the impact of removing partners form the program was never evaluated. The investigators of this study aim to evaluate this.

Therefore, for the MYSLAINTE study, the investigators aim to include patients with stable rheumatoid arthritis and stable 3 or 4 CKD with 2 or more defined uncontrolled cardiovascular risk factors. In order to enter the study, each patient must also have a partner who is willing to take part. Each partner/patient pair will be randomised in a 1:1 ratio into one of two groups: with partner or without partner.

* With partner: the patient and their partner will undergo an initial assessment (week 1), a 10 week intervention program (weeks 2-11) and then an end of program assessment (week 12)
* Without partner: Both the patient and their partner will undergo an initial assessment (week 1) and end of program assessment (week 12) However, only the patient will undergo the 10 week intervention program. The patients partner will receive usual care from their GP.

The intervention phase is part of the MySláinte program and involves, a weekly 1 hour group supervised exercise session, a weekly 1 hour group health promotion workshop, weekly individualised goal setting, weekly individualised exercise prescription and optimisation of cardioprotective medications. This is all run over a 10 week period and delivered in a community setting by a multidisciplinary team including: a physiotherapist, a dietitian, a nurse specialist and physician.

The primary aim of the study is to assess if the 10 week intervention can improve modifiable cardiovascular risk factors in these patients and their partners. A secondary aim of the study is to assess the impact of simultaneously including a partner in this lifestyle intervention program.

ELIGIBILITY:
Inclusion Criteria:

Patients with either stable rheumatoid arthritis OR stable stage 3 or 4 chronic kidney disease with at least 2 uncontrolled cardiovascular risk factors AND a partner who is also willing to take part in the study.

* Stable rheumatoid arthritis (RA). Rheumatoid arthritis as diagnosed by a rheumatologist. Stable meaning that there was no escalation of disease modifying antirheumatic drugs OR escalation in steroid dose/frequency within the previous 6 months. Patients on a stable dose of chronic steroids are eligible for inclusion.
* Stable chronic kidney disease (CKD). CKD can be of any cause. Stable meaning that there was no significant change in renal function over a period of 3 months Stage of CKD is based on the 2012 KDIGO guidelines:19

  * Stage 3 CKD: GFR 30-59ml/min/1.73m2
  * Stage 4 CKD: GFR of 15-29ml/min/1.73m2.

GFR will be calculated based on CKD-EPI equation.

* At least 2 of the 5 following uncontrolled cardiovascular risk factors:
* Hypertension (BP ≥130/80mmHg)
* Active smokers
* BMI ≥30kg/m2
* Dyslipidemia (LDL ≥1.4mmol/L in very high risk, ≥1.8mmol/L with high risk, LDL

  * 2.6mmol/L with moderate risk or ≥3.0mmol/L in low risk)
* Poor glycemic control (Defined as: HbA1c ≥53mmol/mol OR ≥48mmol/mol in patients with a long-life expectancy or type 2 diabetes controlled by diet alone)

All patients with RA/CKD must have a partner to be included in the study. Partners do not need to have any particular underlying diagnosis and can in theory be completely healthy. The partners must not meet any of the exclusion criteria.

Both the patient and the partner must freely sign informed consent.

Exclusion Criteria:

* Known unstable angina, symptomatic severe aortic stenosis, pregnant patients, severe cognitive impairment, physical impairment leading to inability to exercise, currently enrolled in another lifestyle program, currently awaiting organ transplant, previous renal transplant, patients with End Stage Renal Disease (Stage 5 CKD) or those expected to commence dialysis within the next 6 months, acute pulmonary embolus or pulmonary infarction

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2020-03-10 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Improvement in Blood pressure control | 12 weeks
  Blood pressure (systolic) as measured in mmHg
Change in 10 year Cardiovascular Risk score in percent | 12 weeks
  Expressed as a percentage change.
  Calculated using the following link http://www.HeartScore.org
  As all patients will be assessed in Ireland the low risk cardiovascular chart will be used.

SECONDARY OUTCOMES:
Improvement smoking cessation rate | 12 weeks
  Smoking status (self reported smoking status)
  Patients will be asked to report if they are actively smoking at both the initial assessment and the end of program assessment.
Nicotine Dependence | 12 weeks
  This will be assessed using the Fagerstrom score.
  This will be assessed in those who are smoking at the time of the initial assessment and again at the end of program assessment. This score is based on 6 questions and is scored from 0-10. The higher the score, the greater the nicotine dependence.
Improvement in lipid control | 12 weeks
  Lipid Control (Serum total cholesterol, LDL-C, HDL-C and triglycerides)
Improvement in glycaemic control | 12 weeks
  Glycaemic control (serum HbA1c)
Change in body mass index | 12 weeks
  Measured in kilogram per metre squared
Change in waist circumference | 12 weeks
  Measured in centimeters (cm) midway from the lower rib margin to the anterior superior iliac crest while the patient is in the standing position.
Improvement in physical activity levels | 12 weeks
  Physical activity levels (self reported)
  During both the initial assessment and end of program assessment, participants will be asked to record all physical activities that they engaged in for at least 10 minutes at a time over the previous week. They will be asked to further elaborate on the type of activity, approximate duration that they spent doing each activity, how many days they engaged in each activity and a subjective intensity level:
  * Light = felt easy, no shortness of breath
  * Moderate = felt comfortable, makes the patient feel warm, slight out of breath but able to speak a sentence
  * Vigorous = felt hard; felt short of breath and sweaty
Improvement in diet | 12 weeks
  Mediterranean diet score.
  All patients will have a MDS calculated at the time of the initial assessment and then again at the end of program assessment.
  Score ranges from 0-14.
  The higher the score the better the adherence with a Mediterranean diet.
Change in alcohol consumption | 12 weeks
  Self reported alcohol consumption
Change Health assessment questionnaire disability index (HAQ-DI) score | 12 weeks
  Patients with rheumatoid arthritis will be asked to complete the Health assessment questionnaire (HAQ) at the initial assessment and again at the end of program assessment.
  It is a self administered questionnaire.
  This is scored from 0 to 3. The higher the score, the higher the level of disability and the more their underlying condition impacts on their level of daily functioning.
Change in participant reported anxiety | 12 weeks
  Assessed using the Hospital Anxiety and Depression Scale.
  All participants will complete the hospital anxiety and depression scale at the time of the initial assessment and then again at the end of program assessment.
  This is a self administered questionnaire. The higher the score, the higher the level of anxiety.
Change in participant reported depression | 12 weeks
  Assessed using the Hospital Anxiety and Depression Scale.
  All participants will complete the hospital anxiety and depression scale at the time of the initial assessment and then again at the end of program assessment.
  This is a self administered questionnaire. The higher the score, the higher the level of depression.
Change in health related quality of life | 12 weeks
  Assessed using the Dartmouth Primary Care Co-operative functional assessment (COOP)
  A self administered questionnaire. All participants will complete a Darthmouth COOP at the initial assessment and then again at the end of program assessment. The higher the score the worse the participant perceived health related quality of life.
To assess if partners who do not partake in the 10-week intervention phase of the program experience a change in their risk factor profile over the 10-week period by virtue of their partner being involved in the program ("ripple effect") | 12 weeks
  All partners who do not partake in the 10 week intervention phase of the program will have an initial assessment and end of program assessment. They will have all the same indices measured as those partaking in the 10 week intervention as outlined above, which will be used to study the below outcome in these nonparticipating partners:
  Change in 10 year cardiovascular risk score
To assess the adherence of a group of chronic disease patients to a 12-week lifestyle intervention program | 12 weeks
  Adherence to the program will be assessed in all participants with either RA/CKD. A record of the number of sessions attended by each participant will be documented.
  Each patient with CKD/RA will be assigned to attend a total of 12 sessions (an initial assessent, 10 intervention sessions, and then the end of program assessment) The number of these sessions attended will be documented and so they will receive a score out of 12.
To assess the adherence of the partners to a 12-week lifestyle intervention program | 12 weeks
  Adherence to the program will be assessed in all partners. A record of the number of sessions attended by each partner will be documented.
  For partners assigned to the "without partner group" - they will be expected to attend 2 sessions (The initial assessment and end of program assessment) and so will receive a score out of 2.
  For partners assigned to the "with partner" group - they will be expected to attend 12 sessions (the initial assessment, 10 intervention sessions and the end of program assessment) and so will receive a score out of 12.
Change in disease activity score 28-C Reactive Protein (DAS28-CRP) in patients with Rheumatoid Arthritis | 12 weeks
  Patients with Rheumatoid Arthritis will have a Disease Activity Score 28 - CRP calculated at the time of initial assessment and then again at the time of end of program assessment. These two measurements will be compared.
  The DAS28-CRP will provide a number between 0 and 10 to indicate disease activity. Higher numbers indicate more active disease.
Change in urine albumin creatinine ratio (ACR) in patients with chronic kidney disease | 12 weeks
  Those with CKD will have a urine ACR taken at the initial assessment and then again at the end of program assessment. These two measurements will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: John W McEvoy, Principal Investigator — National University of Ireland, Galway
Locations (1):
- Croí, Galway, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gibson I, Flaherty G, Cormican S, Jones J, Kerins C, Walsh AM, Costello C, Windle J, Connolly S, Crowley J. Translating guidelines to practice: findings from a multidisciplinary preventive cardiology programme in the west of Ireland. Eur J Prev Cardiol. 2014 Mar;21(3):366-76. doi: 10.1177/2047487313498831. Epub 2013 Jul 24. PMID 23884981
- See also: Used to calculate a participants estimated cardiovascular risk — http://www.HeartScore.org